CLINICAL TRIAL: NCT04778761
Title: Randomized Trial of a Home-Advance Care Planning Video Intervention for Patients With Life-Limiting Illness
Brief Title: ACP Video Intervention for Patients With Life-Limiting Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Assistant Professor Of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020P001277
Record Dates: First submitted 2021-02-04; First posted 2021-03-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Health Care Utilization; End Stage Disease
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research team collecting study outcomes will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care entails receiving usual medical care by the home-based care team.
- Video intervention (Experimental): In addition to usual care, the intervention will entail having a visit by a trained study clinician to provide access to the ACP video. The study clinician will discuss the content of the video and answer any questions.
  Interventions: Behavioral: Home ACP Video

INTERVENTIONS:
Behavioral: Home ACP Video — A video focused on Advance Care Planning and Hospice for patients with serious illness
  Arms: Video intervention

SUMMARY:
The goal of this research is to increase patients' knowledge about advance care planning (ACP) discussions and hospice care for patients with serious illness receiving home-based care.

DETAILED DESCRIPTION:
ACP is a process that allows patients to communicate their wishes and preferences or medical care, when they are seriously ill, to their medical providers. The study investigators would like to assess whether a home-ACP video can improve patient-clinician communication about patients wishes for their medical care and lead to more patient-centered care.

This study is a randomized clinical trial of a Home-ACP intervention among 500 adult patients with serious illness receiving medical care at home with the Clover Health House Calls Program. Study participants will be assigned to one of two groups. In one group, participants will continue to receive usual care with their home-based care team. In the second group, participants will continue to receive their usual care with their home-based care team and also view an ACP video that helps them understand ACP and provides education about ACP and hospice care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 or over
* Have a one-year prognosis or less as determined by Clover Health's validated algorithm
* Speak either English or one of the other 25 languages in which the video intervention is available

Exclusion Criteria:

* Visually impaired beyond 20/200 corrected
* Acute psychiatric illness or other comorbid condition that impairs cognitive ability to participate in advance care planning discussion as determined by the primary House Call Provider.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospice utilization | up to one year follow-up or death
  Compare the use of hospice (yes vs. no) between the study groups

SECONDARY OUTCOMES:
Hospice length of stay | up to one year follow-up or death
  Compare hospice length-of-stay between the study groups
Rates of documented resuscitation preferences in the Electronic Health Record | up to one year follow-up or death
  Compare documented resuscitation preferences in the Electronic Health Record between the two groups
Rates of Advance Care Planning documentation in the Electronic Health Record | up to one year follow-up or death
  Compare advance care planning documentation in the Electronic Health Record between the two groups
Patient knowledge about Advance Care Planning | Up to two days following the intervention visit
  Compare patient's knowledge about advance care planning using a 5-item knowledge questionnaire (range 0-5), higher score indicate more knowledge
Patient reported confidence in care | up to two days following the intervention visit
  Compare patient's reported confidence in their medical care using a single Likert response question between the two study groups. Score range from 0-4. Higher scores indicate higher confidence in care
Patient reported satisfaction with clinician communication | up to two days following the intervention visit
  Compare patient satisfaction with their communication with their clinician using the CAHPS subscale. Score range 0-20. Higher score indicate better satisfaction with communication
Patient reported decisional satisfaction | up to two days following the intervention visit
  Compare patient reported decisional satisfaction between the study groups using the Satisfaction with Decision Scale. Scale range from 6-30. Higher scores indicate higher satisfaction with decision
Patient reported decisional certainty | up to two days following the intervention visit
  Compare patient reported decisional certainty between the two groups using the Decision Conflict Scale. Score ranges from 0 to 100. Higher scores indicate higher decisional conflict

OTHER OUTCOMES:
Cost of care in the last year of life | 1 year
  Compare cost of care in the last year of life between the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Clover Health, Jersey City, New Jersey, United States